CLINICAL TRIAL: NCT03544333
Title: Boost rTMS for AVH - Therapeutic Response and Neurobiological Prediction Markers in Auditory Verbal Hallucinations
Brief Title: Boost rTMS for Auditory Verbal Hallucinations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of low recruitment numbers.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Philipp Homan, Assistant Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-0024
Record Dates: First submitted 2018-04-27; First posted 2018-06-01 (Actual); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia; Auditory Hallucination
Keywords: transcranial magnetic stimulation (TMS); brain stimulation; medication-free
MeSH Terms: conditions — Schizophrenia; Hallucinations | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- real transcranial magnetic stimulation (Experimental): In the treatment arm, patients will receive 1Hz of repetitive transcranial magnetic stimulation (rTMS) over the left Sylvian parietal temporal area (area Spt) four times on 1 day (1 pulse/second and a total of 1'000 pulses: 16 minutes' protocol at 100 % of motor threshold modified based on Hoffman et al.,1999). Area Spt will be localized via baseline structural imaging and our Localite TMS navigation system.
  Interventions: Device: transcranial magnetic stimulation
- sham transcranial magnetic stimulation (Placebo Comparator): In the comparator arm, patients will receive no stimulation. The TMS coil adjusted to the patients head will not be plugged into the TMS machine and can thus not have an effect on the brain. Yet, patients will hear the same noises from a coil that is plugged in, see the TMS machine running, and area Spt localized via baseline structural imaging and our Localite TMS navigation system.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — We will assess safety and efficacy of the following protocol: 1Hz of rTMS over the Sylvian parietal temporal area (area Spt) four times on 1 day (1 pulse/second and a total of 1'000 pulses: 16 minutes' protocol at 100 % of motor threshold modified based on Hoffman et al., 1999). Area Spt will be localized via baseline structural imaging and our Localite TMS navigation system.

SUMMARY:
This is a randomized, placebo controlled, double-blind clinical trial. The investigators aim to examine the safety and efficacy of repeated transcranial magnetic stimulation (rTMS) for the treatment of auditory verbal hallucinations (AVH) in patients with schizophrenia who are not taking antipsychotic medication. The investigators employ a novel, accelerated protocol with only four sessions of low-frequency rTMS in one day. The effects of this accelerated protocol will be compared to the sham stimulation. Additionally, the investigators will examine the effects of rTMS on a neurophysiological level by evaluating mechanism of action in the temporo-parietal lobe by means of functional magnetic resonance imaging.

DETAILED DESCRIPTION:
Auditory verbal hallucinations affect up to 70% of schizophrenia patients (Waters, 2012), yet, even extended antipsychotic medication does not ameliorate AVH in 20-30% of patients (Sukhwinder S Shergill et al., 2007) and is often accompanied by side effects (Leucht et al., 2009). Therefore, it is crucial to develop and assess promising potentially beneficial therapeutic options.

Non-invasive brain stimulation techniques like repetitive transcranial magnetic stimulation (rTMS) have been proposed to disrupt mechanisms in question. A number of meta-analyses (Aleman, Sommer, & Kahn, 2007; Demeulemeester et al., 2012; Freitas, Fregni, & Pascual-Leone, 2009; C. W. Slotema, Blom, van Lutterveld, Hoek, & Sommer, 2014; C. W. Slotema, Dirk Blom, Hoek, & Sommer, 2010; Tranulis, Sepehry, Galinowski, & Stip, 2008) found significant effect sizes ranging from 0.42 to 1.04 for 1Hz rTMS over the left temporo-parietal junction for the treatment of AVH. However, the majority of studies so far investigated the effects of rTMS in treatment resistant schizophrenia patients as an ad-on or second-line treatment.

No study to date has explored the effects of rTMS either as a first-line treatment or in the initial stage of the illness. This is surprising, considering the fact that rTMS is a safe treatment with minimal side-effects (Rossi, Hallett, Rossini, & Pascual-Leone, 2009) that could be used already in the earlier phase of treatment. This stands in considerable contrast to the range of side-effects associated with antipsychotics (Leucht et al., 2017) that can be disabling for patients and lead to lower quality of life.

Therefore, the crucial next step is (1) to explore the effects of rTMS in medication-free patients from the whole schizophrenia spectrum and (2) to use an accelerated protocol of multiple rTMS-sessions within a short period of time. To make this assessment feasible, considering that patients have to be off medication, the safest and also most efficient way is an accelerated rTMS protocol. The great advantage of such an approach is that the effects of rTMS can be investigated independently of potentially influencing effects of antipsychotics and at the same time assess the efficacy of rTMS within a very short amount of time.

In the proposed study, the investigators aim to determine the efficacy of rTMS as a potential treatment for AVH in schizophrenia and thus reduce suffering in patients and their relatives.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 to 65
4. Diagnosed with Diagnostic and Statistical Manual (DSM) V diagnosis of schizophrenia (295.90), schizoaffective disorder (295.70), or brief psychotic disorder (298.80), prone to AVH in the acute phases of the disorder
5. Willing to adhere to the rTMS regimen
6. No antipsychotic medication in the last two weeks prior to the start of the study as well as no antipsychotic medication during participation in the study
7. Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

1. Current use of antipsychotic medication within the last 2 weeks
2. Electroconvulsive therapy or rTMS within three months (see the TMS screening questionnaire)
3. History of seizures
4. Presence of implanted electronic device or metal implant in the head and neck region (DBS, cochlear implant, etc.)
5. Pregnancy, as assessed with a pregnancy test prior to every MRI measurement, or lactation
6. Any active general medical condition or central nervous system disease which can affect cognition or response to treatment
7. Treatment with another investigational drug or other intervention within 2 weeks
8. Current diagnosis of delirium, dementia, or amnestic amnesiac disorder; Diagnosis of mental retardation; Current (within the past three months) diagnosis of active substance dependence, or active substance abuse within the past week as indicated by self-report.
9. Patients who are cognitively impaired and are thus not able to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Homan, MD PhD, Principal Investigator — Zucker Hillside Hospital, New York City, USA.
Locations (1):
- The Zucker Hillside Hospital, Northwell Health, Manhasset, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Started | 3 | 2
Completed | 2 | 2
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.67 (5.98) | 27.02 (3.75) | 29.84 (5.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
BPRS Total Score [Mean (Full Range); unit: units on a scale] — Brief Psychiatric Rating Scale (BPRS) Note that higher values indicate greater severity: 0 = not assessed, 1 = not present, 2 = very mild, 3 = mild, 4 = moderate, 5 = moderately severe, 6 = severe, 7 = extremely severe.
  The total score is the sum of all 18 items. Population: Pat. did not finish baseline assessment.
  units on a scale
    number analyzed (Participants) | 1 | 2 | 3
    (all) | 36 [31 to 41] | 38 [36 to 40] | 37 [31 to 41]
GAS [Mean (Standard Deviation); unit: units on a scale] — Global Assessment of Functioning (GAF) Note that higher scores indicate more funcitonal impariment: Scores range from 100 (extremely high functioning) to 1 (severely impaired). Population: Patient was not available for assessment.
  units on a scale
    number analyzed (Participants) | 1 | 2 | 3
    (all) | 75 (NA) — Patient was not available for assessment. | 30 (7.07) | 52.5 (NA) — Patient was not available for assessment.
Hallucination Change Score [Mean (Full Range); unit: units on a scale] — Hallucination Change Score (HCS) Note that this scale is centered at 10 (baseline). For the following 3 assessments, participants judges whether the hallucination severity is unchanged (10) has increased (>10 up to 20), has decreased (< 10), or whether they don't hear any hallucinations at all currently (0).
  units on a scale | 7.5 [0 to 15] | 7.5 [5 to 10] | 7.5 [0 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Transcranial Magnetic Stimulation for Auditory Verbal Hallucinations Assessed With the Hallucination Change Scale
Description: Examine change in AVH severity, measured with the Hallucination Change Scale, due to low-frequency rTMS.
  The Hallucination Change Scale is a self-rating assesses severity of hallucinations. It is anchored at baseline using the patient's description of AVH for the previous 24-hours which is assigned a score of 10. The subsequent assessments are in relation to the baseline where a reduction of AVH relates to a value < 10 (best being a value of 0) and a worsening of AVH relates to a value > 10 (twice as severe as baseline being a value of 20).
Time Frame: Four timepoints of the Hallucination Change Scale (after every TMS session). Here, score after final session is reported.
Population: Pat. lost for followup.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Real Transcranial Magnetic Stimulation: In the treatment arm, patients will receive 1Hz of repetitive transcranial magnetic stimulation (rTMS) over the left Sylvian parietal temporal area (area Spt) four times on 1 day (1 pulse/second and a total of 1'000 pulses: 16 minutes' protocol at 100 % of motor threshold modified based on Hoffman et al.,1999). Area Spt will be localized via baseline structural imaging and our Localite TMS navigation system.
  TMS: We will assess safety and efficacy of the following protocol: 1Hz of rTMS over the Sylvian parietal temporal area (area Spt) four times on 1 day (1 pulse/second and a total of 1'000 pulses: 16 minutes' protocol at 100 % of motor threshold modified based on Hoffman et al., 1999). Area Spt will be localized via baseline structural imaging and our Localite TMS navigation system.
- Sham Transcranial Magnetic Stimulation: In the comparator arm, patients will receive no stimulation. The TMS coil adjusted to the patients head will not be plugged into the TMS machine and can thus not have an effect on the brain. Yet, patients will hear the same noises from a coil that is plugged in, see the TMS machine running, and area Spt localized via baseline structural imaging and our Localite TMS navigation system.
  sham stimulation: We will assess safety and efficacy of the following protocol: 1Hz of rTMS over the Sylvian parietal temporal area (area Spt) four times on 1 day (1 pulse/second and a total of 1'000 pulses: 16 minutes' protocol at 100 % of motor threshold modified based on Hoffman et al., 1999). Area Spt will be localized via baseline structural imaging and our Localite TMS navigation system.
Arm/Group | Real Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 2 | 2
score on a scale | 15 [15 to 15] | 7.5 [5 to 10]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the three days.
Description: The definition did not differ.
Groups:
- Real TMS: This group received real TMS.
- Sham TMS: This group received sham TMS.
Arm/Group | Real TMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03544333/Prot_SAP_001.pdf
  • Informed Consent Form (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT03544333/ICF_000.pdf